CLINICAL TRIAL: NCT00838344
Title: The Medication Adherence Program:Promoting Diabetes Self-Management Through Community Pharmacies
Brief Title: The Medication Adherence Program
Acronym: MAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Washington (Other)
Collaborators: American Association of Diabetes Educators (Other)
Responsible Party: Peggy Odegard, Associate Professor, University of Washington
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: 33084-D; 07-9030-D-01; RFA0100-06
Record Dates: First submitted 2009-02-05; First posted 2009-02-06 (Estimated); Last update posted 2009-09-30 (Estimated); Status verified 2009-09

CONDITIONS: Treatment; Diabetes
Keywords: medication adherence; medication persistence; pharmacist interventions; diabetes; persistence; adherence
MeSH Terms: conditions — Diabetes Mellitus; Medication Adherence

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (No Intervention): Usual prescription refill system and pharmacy care.
- Intervention (Experimental): Telephone follow-up call to individuals with diabetes (Type 2) who have missed a prescription refill by 6 or more days. Call includes assessment of refill need, discussion of diabetes care progress and any medication adherence barriers with intervention to resolve barriers.
  Interventions: Other: Medication Adherence Program (MAP)

INTERVENTIONS:
Other: Medication Adherence Program (MAP) — Telephone follow-up call to individuals with diabetes (Type 2) who have missed a prescription refill by 6 or more days. Call includes assessment of refill need, discussion of diabetes care progress and any medication adherence barriers with intervention to resolve barriers.
  Arms: Intervention

SUMMARY:
In this study, the investigators will evaluate the impact of a Medication Adherence Program (MAP), a systematic telephone call to patients who are overdue for refills, to assess individual reasons or barriers to refilling prescribed DM medicines, discuss diabetes care progress, and provide intervention to resolve any barriers to taking prescribed medicines. The hypothesis for the study is that personalized telephone follow-up by a pharmacist will assist people who have missed refilling their prescriptions in taking diabetes medicines by resolving medication adherence challenges. Following randomization, the intervention will be offered to patients of four Seattle-area Safeway Pharmacies, Inc, who are overdue for prescribed DM medicine refills by at least 6 days. Control subjects will receive usual pharmacy care at the participating Safeway pharmacies as a comparison. The study will provide medication adherence support to intervention subjects for 12 months following enrollment with the goal of improving medication refilling and persistence.

DETAILED DESCRIPTION:
Taking medicines can be a challenge for those with diabetes mellitus (DM) with adherence rates to DM medicines as low as 31%. Adherence to DM medicines improves DM by reducing blood glucose (ie A1c reduction) but will also result in improved outcomes, reduced cardiovascular risks, and reduced costs of diabetes. The most common factors reported to affect medication taking in those with DM include difficulty remembering refills and doses, regimen complexity (e.g more than one DM drug, need to split tablets, mix products), dosing frequency greater than twice daily, depression, and adverse effects or fear of them.

Pharmacists have immense opportunity to interact with people with DM, who now number over 20 million in the United States (US). This reality is due to several factors including convenience of pharmacies (found in most urban, suburban, and rural communities), accessibility of pharmacists for questions and counseling (appointments not usually required), and strong rapport that pharmacists and their staff develop with long-term patients and their families through their presence in the community. Pharmacists in community practices work directly with patients and review refill information about patient medication use thus allowing for personalized, immediate, and ongoing promotion of adherence. Currently, pharmacists do not routinely call patients who are overdue for prescription refills to ascertain if the refill is still needed or proactively work to resolve any barriers to refilling. The standard of care is to provide refill and medication adherence support if it is requested by a patient and if the pharmacy is able to provide the needed level of support.

In this study, we will evaluate the impact of a Medication Adherence Program (MAP), a systematic telephone call by a pharmacist to patients who are overdue for refills, to assess individual reasons or barriers to refilling prescribed DM medicines and provide intervention to resolve any barriers.

ELIGIBILITY:
Inclusion Criteria:

* 18 or older with type 2 diabetes on at least one oral diabetes medication who have missed a refill by 6 or more days

Exclusion Criteria:

* Those unable to converse in the same language as their usual care Safeway pharmacist (Spanish or English most common languages spoken at the site stores) or who do not have an interpreter, family member, friend, or caregiver who can act on the subject's behalf as an interpreter during the initial or any follow-up phone calls

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2008-04; Primary Completion 2010-01 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
medication adherence | 12 months

SECONDARY OUTCOMES:
medication adherence challenges | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Washington, Seattle, Washington, United States